CLINICAL TRIAL: NCT06594107
Title: Faktorer För Uppkomst Och Förlopp Av Axial Spondylartrit
Brief Title: Factors for the Onset and Course of Axial Spondylitis
Acronym: EISPA
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Per-Johan Jakobsson, MD PhD Professor, Karolinska Institutet
Other Study IDs: EISPA; 2022-01789-01 (Other: Karolinska Institute and University Hospital)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Axial Spondyloarthritis
Keywords: observational; axial spondyloarthritis; prostaglandins; predictive factors
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Whole blood samples heparin blood, EDTA blood and urine samples are collected at baseline, after 1 and 2 years in the first 100 patients.
  1 group, 2 cohorts 1 at Karolinska and 1 at the center for Rheumatology in Stockholm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1 cohort at Karolinska University Hospital and 1 at the Center for Rheumatology in Stockholm: This cohortstudy is performed at 2 sites.

SUMMARY:
In a research project, investigators want to study the course of the disease of axial spondylitis: the causes of disease onset, prognosis, and treatment effects. The goal is to improve treatment and in the long run also prevention of the disease. The project has a focus on the body's own substance prostaglandin, and its proinflammatory role in spondylitis, but also other substances may be analyzed in blood and urine samples.

The purpose of the research project is include newly diagnosed treatment-naive patients with axial spondyloarthritis, to follow them after 1 and 2 years after treatment start, to collect clinical data, questionnaires, blood and urinsamples to find blood or urine markers that can be used for precision therapy of axial spondylitis.

DETAILED DESCRIPTION:
The EISPA study is an epidemiological and translational study in axial spondylitis patients who are included in the Swedish Rheumatology Quality Register (SRQ). EISPA aims to include consecutive newly diagnosed axial spondylitis patients.

Despite the fact that the disease is relatively common, it takes on average 10 years after start of symptoms for patients be diagnosed with axial spondylitis.

Axial spondylitis diagnosis is based on clinical findings rather than diagnostic tests, which reflects lack of knowledge about what causes the disease. At present, our possibilities to predict the course of the disease (and thereby individualize the care of the patient) are limited. Current treatment decreases inflammation rather than treating the cause of the disease.

The first treatment step of axial spondylitis is with non-steroidal anti-inflammatory drugs or COX inhibitors, which usually have insufficient effect against inflammatory pain and stiffness. In addition, these drugs are associated with side effects, such as gastrointestinal and cardiovascular side effects. Axial spondylitis is a multifactorial disease where the arachidonic acid cascade, an increased prostaglandin production and release may play a major role. With this there is a clear potential to develop new specific drugs to slow down the prostaglandin cascade in patients with axial spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed patients with axial spondyloarthritis
* treatment-naive
* 18 years of age or older
* Swedish-speaking
* Able to give informed consent

Exclusion Criteria:

* DMARD treatment,
* ongoing infection
* ongoing malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive newly diagnosed adult patients with axial spondyloarthritis who are treatment-naïve, speak Swedish, and do not have an ongoing malignancy or infection. Patients need to be able to give an informed consent.
  Investigators include 20 anonymised blood samples of blood donors for comparison of prostaglandin levels.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostaglandin levels | 2 years
  Investigators measure prostaglandin levels in treatment-naïve patients at baseline, and then after therapy start after 1 and 2 years.

SECONDARY OUTCOMES:
Questionnaires | 2 years
  Investigators collect data on modifiable environmental factors and lifestyle that may contribute to the onset of the disease.
Clinical data | 2 years
  Investigators collect clinical data as entered in the Swedish Rheumatology Quality Register (SRQ) plus the ASAS-health index (0-17, with a lower score indicating a better health status), such as inflammatory markers ESR (mm/hour)/CRP (mg/l), and other variables in the ASAS core outcome set for all trials as defined by ASAS-Omeract.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Huddinge, Stockholm County
  - Center for Rheumatology Stockholm, Stockholm, Stockholm County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jakobsson PJ, Thoren S, Morgenstern R, Samuelsson B. Identification of human prostaglandin E synthase: a microsomal, glutathione-dependent, inducible enzyme, constituting a potential novel drug target. Proc Natl Acad Sci U S A. 1999 Jun 22;96(13):7220-5. doi: 10.1073/pnas.96.13.7220. PMID 10377395